CLINICAL TRIAL: NCT06116916
Title: A Phase 2, Multicenter, Randomized, Double-Masked, Parallel-Group Study to Assess the Efficacy and Safety of KHK4951, a Vascular Endothelial Growth Factor Receptor Inhibitor, in Patients With Diabetic Macular Edema
Brief Title: Study to Assess the Efficacy & Safety of KHK4951 in Patients With Diabetic Macular Edema
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4951-003
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Macular Edema (DME)
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): KHK4951 High dose
  Interventions: Drug: KHK4951; Drug: Aflibercept Injection
- Arm B (Experimental): KHK4951 Middle dose
  Interventions: Drug: KHK4951; Drug: Aflibercept Injection
- Arm C (Experimental): KHK4951 Low dose
  Interventions: Drug: KHK4951; Drug: Aflibercept Injection

INTERVENTIONS:
Drug: KHK4951 — KHK4951 eye drop for 36 weeks until end of the trial
Drug: Aflibercept Injection — Intravitreal injection (IVT) of aflibercept will be given as specified in the protocol

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of KHK4951 eye drops in patients with DME.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent to participate in the study
* In Korea, participants must be 19 years or older to be enrolled
* BCVA ETDRS letter score of 78 letters to 35 letters as measured by the ETDRS visual acuity chart in the study eye at screening
* 500 μm ≥ CST ≥ 325 μm in the study eye at screening
* HbA1c ≤ 11% at screening

Exclusion Criteria:

* Any signs of proliferative diabetic retinopathy in the study eye
* History of rubeosis in the study eye
* Uncontrolled glaucoma in the study eye
* Aphakia or pseudophakia with AC-IOL in the study eye
* Active intraocular inflammation in the study eye
* Any current ocular condition for which visual acuity loss would not improve from resolution of macular edema in the study eye
* History of rhegmatogenous retinal detachment in the study eye
* Any current or history of ocular disease other than DME that may confound assessment of the macula or affect central vision in the study eye
* History of the following therapies in the study eye

  * History of vitrectomy surgery, submacular surgery, or other surgical intervention for DME
  * Periocular or intraocular (sub-Tenon or IVT) corticosteroids within 12 weeks prior to Day 1 corticosteroids
  * Previous intraocular device implantation except PC-IOL
  * Laser (any type) to the macular area within 12 weeks prior to Day 1
  * Peripheral retinal photocoagulation therapy within 12 weeks prior to Day 1
  * Previous treatment with IVT anti-VEGF drugs other than ranibizumab, bevacizumab, aflibercept 2 mg, and their biosimilars
  * Treatment with ranibizumab, bevacizumab, aflibercept 2 mg, or their biosimilars within 12 weeks prior to Day 1. Previously treated patients who received these medications more than 12 weeks prior to Day 1 can be enrolled, but the patients should be diagnosed with DME within 3 years prior to Day 1
  * Previous use of Ozurdex® or Iluvien® implant
* Any current or history of endophthalmitis in either eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of 15 or more letters in BCVA (Best corrected visual acuity) as measured by ETDRS visual acuity chart from baseline | For 36 weeks until the end of the trial

SECONDARY OUTCOMES:
The number of aflibercept IVT | For 36 weeks until the end of the trial
Change from baseline in SHRM as measured by SD-OCT | 36 Weeks
Change from baseline in retinal morphology as measured by SD-OCT | 36 Weeks
Change from baseline in leakage as measured by FA | 36 Weeks

OTHER OUTCOMES:
Number of participants with adverse events | For 36 weeks until the end of the trial
Serum KHK4951 concentration | 36 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sotaro Takigawa, Study Director — Kyowa Kirin Co., Ltd.
Locations (87):
- United States (40):
  - Barnet Dulaney Perkins Eye Center - Phoenix, Mesa, Arizona
  - Retina Associates Southwest, P.C., Tucson, Arizona
  - Win Retina, Arcadia, California
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - The Retina Partners, Encino, California
  - Salehi Retina Institute, Inc, Huntington Beach, California
  - California Eye Specialists Medical Group Inc, Pasadena, California
  - Retina Consultants of Southern California, Redlands, California
  - Retina Consultants of Southern CO, Colorado Springs, Colorado
  - Blue Ocean Clinical Research West, Clearwater, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Eye Associates of Pinellas, Pinellas Park, Florida
  - Ft. Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Associates of Florida - Saint Petersburg, St. Petersburg, Florida
  - Southern Vitreoretinal Associates, Tallahassee, Florida
  - Center for Retina and Macular Disease - Ophthalmology, Winter Haven, Florida
  - Mid Atlantic Retina Specialists - Hagerstown, Hagerstown, Maryland
  - Sierra Eye Associates, Reno, Nevada
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Vision Research Center Eye Associates of New Mexico, Albuquerque, New Mexico
  - Retina Vitreous Surgeons of Central NY, PC, Liverpool, New York
  - Ophthalmic Consultants of Long Island, Oceanside, New York
  - Retina Vitreous Center in Edmond Oklahoma, Edmond, Oklahoma
  - EyeHealth Northwest, Portland, Oregon
  - Wills Eye Health System, Bethlehem, Pennsylvania
  - Eye Care Specialists, Kingston, Pennsylvania
  - Retina Consultants of Charleston - (RCA Network Site), Charleston, South Carolina
  - Charleston Neuroscience Institute (RCA Network Site), Ladson, South Carolina
  - Black Hills Regional Eye Institute - Ophthalmology, Rapid City, South Dakota
  - Charles Retina Institute, Germantown, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Retina Associates - Ophthalmology/Retina (RCA Network site), Austin, Texas
  - Austin Clinical Research, LLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Retinal Consultants of Texas- San Antonio (RCA Network site), San Antonio, Texas
  - Retina Consultants of Texas (RCA Network Site), The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - University of Vermont Fletcher Allen Health Care, Burlington, Vermont
  - Retina Group of Washington, Fairfax, Virginia
- Australia (9):
  - Eye Clinic Albury Wodonga, Albury, New South Wales
  - South West Retina, Liverpool, New South Wales
  - Marsden Eye Specialists, Parramatta, New South Wales
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic & Day Surgery, Sydney, New South Wales
  - Adelaide Eye and Retina Centre, Adelaide, South Australia
  - Hobart Eye Surgeons, Hobart, Tasmania
  - Centre for Eye Research Australia, East Melbourne, Victoria
- Japan (24):
  - Aichi Medical University Hospital - Ophthalmology, Nagakute, Aichi-ken
  - MIYAKE Eye Hospital, Nagoya, Aichi-ken
  - Toho University Medical Center Sakura Hospital, Sakura, Chiba
  - Kurume University Hospital, Kurume, Fukuoka
  - Minamitohoku Eye Clinic, Kōriyama, Fukushima
  - Caress Sapporo Tokeidai Memorial Hospital, Sapporo, Hokkaidô
  - Kobe University Hospital - Ophthalmology, Kobe, Hyôgo
  - Kozawa Eye Hospital and Diabetes Center, Mito, Ibaraki
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Shinshu University Hospital - Ophthalmology, Matsumoto, Nagano
  - Nara Medical University Hospital - Ophthalmology, Kashihara, Nara
  - Kansai Medical University Medical Center, Hirakata, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Muramatsu Clinic Muramatsu Eye Clinic - Ophthalmology, Susono, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Nihon University Hospital, Chiyoda City, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Hachiōji, Tokyo
  - Tokyo Medical Center, Meguro City, Tokyo
  - Keio University Hospital - Ophthalmology, Shinjuku, Tokyo
  - Hayashi Eye Hospital - Ophthalmology, Fukuoka
  - Fukushima Medical University Hospital - Ophthalmology, Fukushima
  - Rakuwakai Otowa Hospital, Kyoto
  - Saitama Red Cross Hospital, Saitama
  - Osaka Metropolitan University Hospital, Osaka, Ôsaka
- South Korea (14):
  - Keimyung University Dongsan Hospital, Daegu, Dalseo-gu
  - Pusan National University Hospital, Busan, Gudeok-ro
  - Seoul National University Bundang Hospital, Seongam, Gyeonggido
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggido
  - Yeungnam University Hospital, Daegu, Nam-gu
  - Gachon University Gil Medical Center, Incheon, Namdong-gu
  - Korea University Anam Hospital, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - Kim Eye hospital, Seoul, Seoul Teugbyeolsi
  - Kyung Hee University Hospital, Seoul, Seoul Teugbyeolsi
  - The Catholic Univ of KOR, SSMH, Seoul

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the study sponsored by Kyowa Kirin will be available in the Vivli repository, https://vivli.org/ourmember/kyowakirin/ as long as conditions of data disclosure specified in the policy section of the Vivli website are satisfied.